CLINICAL TRIAL: NCT06943924
Title: COMPARISON OF CCI, EmSFI AND fTRST SCORING SYSTEMS IN PREDICTION OF MORTALITY IN EMERGENCY GENERAL SURGERY CASES OVER 65 YEARS OF AGE
Brief Title: A Comparative Study of CCI, EmSFI, and FTRST Scoring Systems
Status: Completed | Type: Observational
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, GUHER TUNA DELIKANLI, assistant doctor of anesthesiology, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Other Study IDs: GDELIKANLI; 010.99/16 (Other: Dr Lutfi Kirdar City Hospital)
Record Dates: First submitted 2025-04-17; First posted 2025-04-25 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: One Hundred Patients Aged 65 and Older Who Underwent Emergency General Surgical Interventions; Clinical Utility of These Scoring Systems; Gastrointestinal Neoplasms; Appendicitis Acute; Emergency Surgery Patients
Keywords: Emergency surgery; Frailty assessment; Mortality prediction
MeSH Terms: conditions — Gastrointestinal Neoplasms; Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Frailty assessment — This study aims to investigate the accuracy and clinical utility of these scoring systems in predicting mortality in individuals aged 65 and older undergoing emergency surgery.

SUMMARY:
Frailty assessment tools and comorbidity indices play a crucial role, particularly in predicting outcomes for elderly patients undergoing emergency surgery. The Emergency Surgery Frailty Index (EmSFI), Charlson Comorbidity Index (CCI), and the Flemish version of the Triage Risk Screening Tool (fTRST) are considered valuable tools that help understand patients perioperative risk profiles. This study aims to investigate the accuracy and clinical utility of these scoring systems in predicting mortality in individuals aged 65 and older undergoing emergency surgery

ELIGIBILITY:
Inclusion Criteria Patients aged 65 years and older who underwent emergency abdominal surgery

Exclusion Criteria:

* Multiple hospitalizations for the same pathology,
* Initial admission at another facility,
* History of emergency abdominal surgery before the study period,
* Terminal-stage cancer
* Emergency reoperations following elective surgery,
* Surgery while in the intensive care unit.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 65 years and older who underwent emergency abdominal surgery .
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-10-23 (Actual)

PRIMARY OUTCOMES:
Predicting 30-Day Mortality in Elderly Emergency Surgery Patients: A Comparative Study of CCI, EmSFI, and fTRST Scoring Systems | From enrollment to the postoperative at 1 month
  This study aims to investigate the accuracy and clinical utility of these scoring systems in predicting mortality in individuals aged 65 and older undergoing emergency surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Lutfi Kirdar City Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided